CLINICAL TRIAL: NCT04652713
Title: Breakfast for Young Women
Acronym: GoDag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: P11-GoDag
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Wolman Disease; Nutrition
MeSH Terms: conditions — Obesity; Wolman Disease

STUDY DESIGN:
Intervention Model Description: Single-blind randomized crossover trail with three intervention meals.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High protein breakfast (Experimental): Participants will be served a dairy-based protein-rich breakfast meal.
  Interventions: Other: Protein-rich breakfast
- High carbohydrate breakfast (Experimental): Participants will be served a carbohydrate-rich breakfast meal
  Interventions: Other: Carbohydrate-rich breakfast
- No breakfast (Experimental): Participants will be served no breakfast
  Interventions: Other: No breakfast

INTERVENTIONS:
Other: Protein-rich breakfast — High protein yoghurt containing approx. 10 g protein per 100 g. Participants will be asked to consume 300 g (=3 dl) yoghurt with 40 g oats for breakfast.
  1 glas of water (150 ml)
  Arms: High protein breakfast
Other: Carbohydrate-rich breakfast — Low protein breakfast containing approx. 2 g protein per 100 g. Participants will be asked to consume ~60 g bread, 20 g jam and 250 ml juice for breakfast.
  1 glas of water (150 ml)
  Arms: High carbohydrate breakfast
Other: No breakfast — 1 glas of water (150 ml)
  Arms: No breakfast

SUMMARY:
Investigators will in a crossover study test the health effects of eating a dairy-based protein-rich breakfast, isocaloric carbohydrate-rich breakfast or no breakfast in young overweight women. Determination of satiety and hunger using visual analog scores (VAS), collection of blood samples and 2x 24 hours food logs will be collected.

DETAILED DESCRIPTION:
This study is a single-blind randomized Cross-Over trial with 30 women aged 18-30 years, each completing three trials. Participants will consume either dairy-based protein-rich breakfast, isocaloric, fiber matched, fat matched, carbohydrate-rich breakfast or no breakfast in randomized order. Three hours later a standardized ad libitum lunch will be served.

Blood samples will be collected (pre, 10 min, 30 min, 60 min, 120 min, 175 min after breakfast) and VAS rating hunger, satiety and desire to eat will be determined (pre, during breakfast, 10, 30, 60, 90, 120, 180 min, during lunch, after lunch). Twenty-four hour food logs on the day before the test day and on the test day will be collected.

Participants will be characterized by determining height (cm), weight (kg), and body composition by a dual-energy X-ray (DXA) scan before the first test day.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 25
* Age 18-25 years
* Regular exercise < 5 hour per week

Exclusion Criteria:

* illness and use of medication affecting the study outcomes
* allergy towards lactose or gluten
* weightloss/gain >5kg the last 6 months
* dieting
* eating disorder
* pregnancy
* breast feeding
* unable to speak and understand danish

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Energy consumption on test days | 0-24 hours
  Total energy consumption on test days (24 hour food log)

SECONDARY OUTCOMES:
Change in hunger | 0-3 hours
  Visual Analog Scale (10 cm) score for feeling of hunger
Change in satiety | 0-3 hours
  Visual Analog Scale (10 cm) score for feeling of satiety
change in desire | 0-3 hours
  Visual Analog Scale (10 cm) score for feeling of desire to eat
Change in ghrelin | 0-3 hours
  in blood sample
Change in leptin | 0-3 hours
  in blood sample
Change in glucose-dependent insulinotropic polypeptide (GIP) | 0-3 hours
  in blood sample
Change in Peptide YY (PYY3-36) | 0-3 hours
  in blood sample
Change in insulin | 0-3 hours
  in blood sample
Change in glucagon | 0-3 hours
  in blood sample
Change in glucose | 0-3 hours
  in blood sample
Energy consumption the day before a test day (food registration) | 0-24 hours
  Total energy consumption on the day before the test day

OTHER OUTCOMES:
Height | Baseline
  Height in cm
Weight | Baseline
  Weight in kg
Body composition fat | Baseline
  DXA-scanning to determine fat mass
Body composition fat free | Baseline
  DXA-scanning to determine fat free mass

CONTACTS AND LOCATIONS:
Overall Officials: Mette Hansen, Assoc Prof, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Department for Public Health, Section for Sport Science, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No